CLINICAL TRIAL: NCT06528782
Title: The Effect of Antenatal Breastfeeding Education Given by Pecha Kucha Method on Postpartum Breastfeeding Self-Efficacy, Infant Feeding Attitude and Breastfeeding Satisfaction: a Randomized Controlled Study
Brief Title: The Effect of Breastfeeding Education Given by Pecha Kucha Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Filiz Ünal Toprak, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SBU-EBE-ZB-02
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Breast Feeding
Keywords: Breast Feeding; Midwifery; Breast Feeding Education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Two groups with pecha kucha group and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the application will be performed by the researcher, patients will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pecha Kucha Group (Experimental): Pregnant women who meet the inclusion criteria assigned to the Pecha Kucha group will be informed about the study and their written and verbal consent will be obtained. Pregnant women will be asked to fill out the 'Introductory Characteristics Information Form', the 'Antenatal Breastfeeding Self-Efficacy Scale Short Form' and the 'Infant Feeding Attitude Scale (IOWA)' before the training at the first encounter, and then breastfeeding training prepared by the Pecha Kucha method will be given. 2 weeks after the training, she will be followed up by phone and asked to answer the Pospartum Breastfeeding Self-Efficacy Scale Short Form, Infant Feeding Attitude Scale (IOWA) and Visual Comparison Scale Satisfaction (VAS-M) scale. 4 weeks after the training, she will be asked to answer the Pospartum Breastfeeding Self-Efficacy Scale Short Form, Infant Feeding Attitude Scale (IOWA) and Visual Comparison Scale Satisfaction (VAS-M) scale.
  Interventions: Other: Pecha Kucha method
- Control Group (No Intervention): Pregnant women who meet the inclusion criteria and who are assigned to the control group will be informed about the study and their written and verbal consent will be obtained. Pregnant women will be asked to fill out the 'Descriptive Characteristics Information Form', 'Antenatal Breastfeeding Self-Efficacy Scale Short Form' and 'Infant Feeding Attitude Scale (IOWA)' at the first encounter. After 2 weeks, she will be followed up by telephone and asked to answer the Pospartum Breastfeeding Self-Efficacy Scale Short Form, Infant Feeding Attitude Scale (IOWA) and Visual Comparison Scale Satisfaction (VAS-M). After 4 weeks, she will be asked to answer the Pospartum Breastfeeding Self-Efficacy Scale Short Form, Infant Feeding Attitude Scale (IOWA) and Visual Comparison Scale Satisfaction (VAS-M).

INTERVENTIONS:
Other: Pecha Kucha method — The Pecha Kucha method will be prepared in the form of a presentation consisting of 20 slides each shown for 20 seconds. The Pecha Kucha presentation lasts 6 minutes and 40 seconds, and most slides present only images. This method is planned to be used in breastfeeding education as it will be more memorable because it contains more visual, auditory and short information.
  Arms: Pecha Kucha Group

SUMMARY:
To evaluate the effect of breastfeeding education given with Pecha Kucha method in the prenatal period on breastfeeding self-efficacy, infant feeding attitude and breastfeeding satisfaction in the postpartum period.

DETAILED DESCRIPTION:
Breastfeeding is the most important factor in infant nutrition. Breast milk is a nutritional source that contains the necessary nutrients for the healthy growth of infants after birth and has many benefits in terms of growth and development. However, although the rate of breastfeeding has increased today compared to the past, it is still not at the desired level. In order to increase breastfeeding rates, breastfeeding trainings should be given starting from the prenatal period. In this study, breastfeeding training will be given to pregnant women with pecha kucha method in the prenatal period and the effect of breastfeeding training on postpartum breastfeeding self-efficacy, infant feeding attitude and breastfeeding satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the research,
* To be able to speak and understand Turkish,
* Over 18 years of age,
* At least primary school graduate,
* Gestational week 38 weeks and above
* No chronic illness,
* Pregnant women without communication barriers will be included in the study.

Exclusion Criteria:

* Have a medical indication that prevents breastfeeding,
* Multiple pregnancies,
* A person with a mental illness,
* Not wanting to continue the research process,
* The one who still hasn't given birth 2 weeks after the training,
* Not having their baby with them after childbirth,
* Pregnant women who cannot be reached during the follow-up period will be excluded from the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women 38 weeks and over
Enrollment: 75 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Antenatal and Pospartum Breastfeeding Self-Efficacy Scale Short Form | 0,2 and 4 weeks
  The scale can be administered in prenatal and postnatal periods and measures how competent women feel about breastfeeding. The items of the five-point Likert-type scale are scored as not at all sure, not very sure, sometimes sure, sure, very sure. The lowest score that can be obtained from all the evaluation scores of the scale is 14 and the highest score is 70. A low total score on the scale indicates a low perception of breastfeeding self-efficacy. In the original scale, the Cronbach's alpha reliability coefficient of the prenatal form was 0.87 and the Cronbach's alpha reliability coefficient of the postnatal form was 0.86.

SECONDARY OUTCOMES:
Infant Feeding Attitude Scale (IOWA) | 0,2 and 4 weeks
  Women's attitudes towards breastfeeding and to predict breastfeeding duration as well as the choice of infant feeding method. The scale consists of 17 items on a 5-point Likert scale ranging from (strongly disagree) to (strongly agree). While 9 items in the scale are positive about breastfeeding, 8 items contain positive statements about formula feeding. Formula feeding items are reverse scored. The total attitude score ranged from 17 points (reflecting a positive attitude towards bottle feeding) to 85 points (reflecting a positive attitude towards breastfeeding). Cronbach Alpha internal consistency coefficient was 0.71 and the scale was found to be reliable.
Visual Assessment Scale - Satisfaction (VAS - S) | 2 and 4 weeks
  The VAS is also used to measure other components besides pain, such as satisfaction.In our study, the VAS will also be used to assess mothers' breastfeeding satisfaction levels. The Visual Assessment Scale - Satisfaction (VAS-S) is a 10 cm ruler with the expression "Not satisfied" on one end and "Very satisfied" on the other end. The mother is asked to rate her satisfaction with breastfeeding after the training from 1 to 10. High scores on the scale indicate that the satisfaction of the recipients is also high.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Bicav, Principal Investigator — Saglik Bilimleri Universitesi; Filiz Ünal Toprak, PhD, Principal Investigator — Saglik Bilimleri Universitesi; Ceren Ceyda İşbuğa, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No